CLINICAL TRIAL: NCT03770897
Title: Laparoscopic Appendectomy Performed by Junior SUrgeonS: Impact of 3D Visualization on Surgical Outcome. Randomized Multicenter Clinical Trial
Brief Title: Laparoscopic Appendectomy Performed by Junior SUrgeonS: Impact of 3D Visualization on Surgical Outcome
Acronym: LAPSUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Nereo Vettoretto, Head of Surgery, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NVettoretto
Record Dates: First submitted 2018-08-28; First posted 2018-12-10 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Appendicolith; Appendicitis; Appendicitis With Perforation; Appendicitis Peritonitis; Appendiceal Abscess; Appendicitis Acute
Keywords: 3d Laparoscopy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D laparoscopic appendectomy. (Experimental): Laparoscopic appendectomy will be performed with 3d technology device by young surgeons, tutored by an expert assistant.
  Interventions: Procedure: 3D Laparoscopic Appendectomy
- 2D laparoscopic appendectomy. (Active Comparator): Laparoscopic appendectomy will be performed by young surgeons (tutored by an expert assistant) with the standard 2D viewing method.
  Interventions: Procedure: 2D Laparoscopic Appendectomy

INTERVENTIONS:
Procedure: 3D Laparoscopic Appendectomy — surgical removal of inflamed cecal appendix by 3D laparoscopic procedure
  Arms: 3D laparoscopic appendectomy.
Procedure: 2D Laparoscopic Appendectomy — surgical removal of inflamed cecal appendix by 2D laparoscopic procedure
  Arms: 2D laparoscopic appendectomy.

SUMMARY:
Laparoscopy has revolutionized the approach to a number of surgical problems causing a re-evaluation of several clinical strategies. Now it has become the standard treatment for majority of ailments including symptomatic gall stone disease, appendicitis, GERD (gastroesophageal reflux disease), morbid obesity and colorectal disease. All these developments aim at minimizing perioperative morbidities, providing rapid postoperative recovery and enhancing patient's safety profile. One of the major limitations of conventional laparoscopy is lack of depth perception. Introduction of 3D imaging, has removed many of these technical obstacles. In 1993, Becker et al., reported that a 3D display might improve laparoscopic skills. Since then, many researchers have demonstrated benefit of 3D imaging . Starting from this, we can theorize an impact of 3D technologies on surgeon's learning curves. This concern is recently being demonstrated in experimental and clinical setting with improvement of hand-eye coordination, better laparoscopic skills and less time to learn surgical procedure. Usually junior surgeons (JS) start their activities with cholecystectomy and appendectomy but, despite an amount of literature regarding the first procedure, there is a 'black hole' regarding the use of 3D imaging in laparoscopic appendectomy (LA).

The investigators decided to investigate the impact of 3D visualization on surgeons' and surgical outcome during laparoscopic appendectomy (LA) performed by junior surgeons (JS). Operative details and clinical aspect are both take in account in order to looking for any advantages or concerns conferred on JS in performing LA.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled to undergo laparoscopic appendectomy. Ages eligible for study: >18 Sexes eligible for study: All

Exclusion Criteria:

* Patients who decline to join the study
* Patients under 18 years old
* Patients with contraindication to undergo laparoscopic surgery.
* Patients without appendicular disease found at laparoscopy (such as complicated inflammatory bowel disease, tumor, complicated diverticula, gynecological disorder)
* Patients undergoing open appendectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Operative time. | 1 minute after surgery
  Time taken for the completion of the procedure

SECONDARY OUTCOMES:
Conversion to open appendectomy. | 1 minute after surgery
  Compare the rate of conversion between each arm.
Intraoperative complication | 1 minute after surgery
  Accidental bowel or bladder perforation, uncontrolled bleeding.
Post-operative complication. morbidity, readmission at 30th days, mortality | 30 days
  Post-operative complication. morbidity, readmission at 30th days, mortality
Surgeon's comfort | 1 hour after surgery
  based on questionnaire following the operation: LIKERT scale: from 1 to 5 points for 8 items divided in 2 evaluation: surgical outcome and surgical strain.
  Surgical outcome:
  item 1: surgical skill perception item 2: definition of surgical field item 3: deep perception
  Surgical strain:
  item1: hand and wrist strain item 2: neck strain item 3: back strain item 4: eye strain item 5: performance anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Presidio Ospedaliero di Montichiari, ASST degli Spedali Civili di Brescia, Montichiari, Brescia, Italy